CLINICAL TRIAL: NCT00888706
Title: Effect of Activities and Exercise on Sleep in Dementia
Brief Title: Effect of Activities and Exercise on Sleep in Elderly Persons With Dementia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Dr. Kathy C. Richards, Polisher Research Institute; Abramson Center for Jewish Life
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: R01NR007771 (NIH); R01NR007771 (NIH)
Record Dates: First submitted 2009-04-24; First posted 2009-04-28 (Estimated); Last update posted 2009-04-28 (Estimated); Status verified 2009-04

CONDITIONS: Dementia; Elderly; Sleep
MeSH Terms: conditions — Dementia | interventions — Walking

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Active Comparator)
  Interventions: Behavioral: Control Condition
- 2 (Active Comparator)
  Interventions: Behavioral: Individualized Social Activities (ISA)
- 3 (Active Comparator)
  Interventions: Behavioral: Physical Resistance Training and Walking (PRT/walking)
- 4 (Experimental)
  Interventions: Behavioral: Combined ISA/PRT/walking

INTERVENTIONS:
Behavioral: Control Condition — The group participated in the usual nursing home activities and routines.
  Arms: 1
Behavioral: Individualized Social Activities (ISA) — The group received individualized social activities one hour daily, during usual brief daytime napping episodes, between 9 am to 5 pm in brief 15-30 minute intervals five days a week.
  Arms: 2
Behavioral: Physical Resistance Training and Walking (PRT/walking) — The group participated in high intensity PRT to the hip and arm extensors (three sets of eight repetitions per muscle per group, approximately 40 minutes) plus 10 minutes of warm-up and 10 minutes of cool-down on Monday, Wednesday and Friday afternoons for one hour (between 2-5pm). On Tuesdays and Thursdays, participants walked with a research assistant for as long as the participant could walk for up to 60 minutes.
  Arms: 3
Behavioral: Combined ISA/PRT/walking — The group had one hour of ISA in the morning or afternoon and one hour of PRT/walking in the afternoon from 2-5pm five days a week. This group received interventions for 2 hours per day.
  Arms: 4

SUMMARY:
The purpose of the study is to determine whether individualized social activities, physical resistance training and walking, and a combination of both are effective in improving nighttime sleep in elders with dementia.

DETAILED DESCRIPTION:
Elders with cognitive impairment usually do not a get a good night's sleep and wake up often during their sleep at night. Increased daytime individualized social activity and physical resistance training with walking have the potential to increase nighttime sleep in elders. This can lead to a better quality of life, a decrease in caregiver burden and decrease in nighttime falls for this population and associated fiscal savings.

Consent forms for this RCT, were written in large print, followed all the guidelines of the Institutional Review Board of the University of Arkansas for Medical Sciences, and assured the participants that their participation in the study was voluntary.

ELIGIBILITY:
Inclusion Criteria:

* Age 55 years old or older
* Mini Mental State Examination (MMSE)of 4-26, indicating dementia or mild cognitive impairment
* Less than seven hours of nocturnal sleep and 30 minutes of daytime sleep
* At least two weeks residency in the nursing home
* Medical diagnosis of dementia; AND
* Ability to stand with assistance

Exclusion Criteria:

* Documented near-terminal or unstable medical conditions
* Unresolved malignancy
* Treatment with chemotherapy; AND
* Unstable cardiovascular disease

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 355 (Actual)
Dates: Start 2002-08; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Total sleep time at night and amplitude of the sleep wake rhythm. | 7 weeks

SECONDARY OUTCOMES:
To explore the roles of daytime napping, muscle strength, and physical activity for mediating the effect of Physical Resistance Training (PRT) and walking on total sleep time at night. | 7 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Little Rock, Arkansas, United States

REFERENCES:
- [Background] Richards K, Shue VM, Beck CK, Lambert CW, Bliwise DL. Restless legs syndrome risk factors, behaviors, and diagnoses in persons with early to moderate dementia and sleep disturbance. Behav Sleep Med. 2010;8(1):48-61. doi: 10.1080/15402000903425769. PMID 20043249
- [Background] Richards KC, Roberson PK, Simpson K, Lambert CW, Bliwise DL, Cole CS, Enderlin C, Shue VM, Siddiqui N, Williams JS. Periodic leg movements predict total sleep time in persons with cognitive impairment and sleep disturbance. Sleep. 2008 Feb;31(2):224-30. doi: 10.1093/sleep/31.2.224. PMID 18274270
- [Derived] Herrick JE, Puri S, Richards KC. Resistance training does not alter same-day sleep architecture in institutionalized older adults. J Sleep Res. 2018 Aug;27(4):e12590. doi: 10.1111/jsr.12590. Epub 2017 Aug 10. PMID 28795452
- [Derived] Herrick JE, Bliwise DL, Puri S, Rogers S, Richards KC. Strength training and light physical activity reduces the apnea-hypopnea index in institutionalized older adults. J Am Med Dir Assoc. 2014;15(11):844-6. doi: 10.1016/j.jamda.2014.08.006. Epub 2014 Oct 5. PMID 25294621
- [Derived] Lorenz RA, Gooneratne N, Cole CS, Kleban MH, Kalra GK, Richards KC. Exercise and social activity improve everyday function in long-term care residents. Am J Geriatr Psychiatry. 2012 Jun;20(6):468-76. doi: 10.1097/JGP.0b013e318246b807. PMID 22617163
- [Derived] Richards KC, Lambert C, Beck CK, Bliwise DL, Evans WJ, Kalra GK, Kleban MH, Lorenz R, Rose K, Gooneratne NS, Sullivan DH. Strength training, walking, and social activity improve sleep in nursing home and assisted living residents: randomized controlled trial. J Am Geriatr Soc. 2011 Feb;59(2):214-23. doi: 10.1111/j.1532-5415.2010.03246.x. PMID 21314643